CLINICAL TRIAL: NCT01011101
Title: Internal Monitoring of Eye Movement in Schizophrenia
Status: Terminated | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 100016; 10-EI-0016
Record Dates: First submitted 2009-11-10; First posted 2009-11-11 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2016-08-16

CONDITIONS: Schizophrenia
Keywords: Saccadic Eye Movements; Schizophrenia; Healthy Volunteer; HV
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
Background:

* Researchers are studying how humans are able to move our eyes to a remembered region even when the target has disappeared. The ability to do this suggests that the brain can keep track of where the eyes have looked, without an external target for continued reference. This is called corollary discharge.
* Other research has indicated that patients with schizophrenia might have difficulty monitoring their eye movements. The corollary discharge process may be defective in patients with schizophrenia, and perhaps delayed in time. Researchers have developed a test to examine this possibility in the hope of learning more about schizophrenia and eye movement.

Objectives:

- To assess whether there is a defect in internal monitoring of eye movements in patients with schizophrenia.

Eligibility:

* Individuals over 18 years of age who are able to give informed consent and are able to concentrate on a 20-minute task that involves following projected targets and moving their eyes to remembered locations.
* Individuals with schizophrenia will be recruited from an ongoing NIH protocol studying schizophrenia.
* In addition healthy will be recruited for this protocol.

Design:

* Researchers will check participants' vision in each eye, and ask them to sit at a machine that measures eye movement in order to complete research tasks. Researchers will monitor participants ability to complete these tasks.
* The first task involves simply following a target that jumps to different parts of the screen.
* The second is a 2-step task, in which a participant is asked to look at two separate light targets and then look at the remembered target positions when the lights are off.
* This protocol does not provide treatment. Participants will remain under the care of their own physicians during participation in this protocol.

DETAILED DESCRIPTION:
OBJECTIVE:

To study if there is a defect in internal monitoring of eye movements in patients with schizophrenia.

STUDY POPULATION:

Patients with schizophrenia and normal controls.

DESIGN:

Patients and controls will be asked to follow targets to remembered locations and their eye movements will be monitored.

OUTCOME MEASURES:

Eye movements will be examined for evidence of internal monitoring (corollary discharge) defects which would result in mislocalizing remembered targets.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Adult subjects over 18 years of age who are able to give informed consent and are able to concentrate on a task for 20 minutes which involves following projected targets and moving their eyes to remembered locations.

EXCLUSION CRITERIA:<TAB>

1. Large refractive error requiring strong glasses. Glasses may interfere with the video eye movement recording system. However, participants may wear contact lenses. Subjects with a history of eye disease affecting vision or eye movements will also be excluded.
2. Participants with guardians will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2009-11-02; Study Completion 2016-08-16

PRIMARY OUTCOMES:
Comparison of recordings between groups | End of study

CONTACTS AND LOCATIONS:
Overall Officials: Edmond J FitzGibbon, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Andreasen NC, Nopoulos P, O'Leary DS, Miller DD, Wassink T, Flaum M. Defining the phenotype of schizophrenia: cognitive dysmetria and its neural mechanisms. Biol Psychiatry. 1999 Oct 1;46(7):908-20. doi: 10.1016/s0006-3223(99)00152-3. PMID 10509174
- [Background] Campanella S, Guerit JM. How clinical neurophysiology may contribute to the understanding of a psychiatric disease such as schizophrenia. Neurophysiol Clin. 2009 Feb;39(1):31-9. doi: 10.1016/j.neucli.2008.12.002. Epub 2009 Jan 9. PMID 19268845
- [Background] Duhamel JR, Goldberg ME, Fitzgibbon EJ, Sirigu A, Grafman J. Saccadic dysmetria in a patient with a right frontoparietal lesion. The importance of corollary discharge for accurate spatial behaviour. Brain. 1992 Oct;115 ( Pt 5):1387-402. doi: 10.1093/brain/115.5.1387. PMID 1422794